CLINICAL TRIAL: NCT00291954
Title: A Multicentric, Randomised Study Comparing the Immunogenicity and Safety of Henogen's Adjuvanted Hepatitis B Vaccine Given at 0, 1months to That of Aventis Pasteur MSD's Hepatitis B Given at 0, 1 Months in Pre-Dialysis, and Dialysis Patients Did Not Respond to Previous Hepatitis B Vaccination
Brief Title: Compare the Immune Response & Safety Elicited by Henogen's Adjuvanted Hepatitis B Vaccine vs Aventis Pasteur MSD's Hepatitis B Vaccine in Pre-Dialysis & Dialysis Patients Who Did Not Respond to Previous Hepatitis B Vaccination
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Henogen (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sophie Houard CSO, Henogen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HN017/HBV-003 (105762); NCT00671762 (obsolete NCT alias)
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2008-08-28 (Estimated); Status verified 2008-08

CONDITIONS: Hepatitis B
Keywords: Dialysis; Pre-dialysis; Hepatitis B vaccine; Prophylaxis hepatitis B infection
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Henogen hepatitis B vaccine
  Interventions: Biological: HB-AS02V
- 2 (Active Comparator): HBVAXPRO hepatitis B vaccine
  Interventions: Biological: HBVAXPRO vaccine

INTERVENTIONS:
Biological: HB-AS02V — HB-AS02V (20µg HBsAg) will be administered at Month 0 and 1
  Arms: 1
Biological: HBVAXPRO vaccine — HBVAXPRO vaccine (40µg HBsAg) will be administered at Month 0 and 1
  Arms: 2

SUMMARY:
Hepatitis B prevention in non-responders uraemic patients is currently based on both HBsAg surveillance and the isolation from HBsAg carriers. A more immunogenic vaccine would be a benefit for this population.

DETAILED DESCRIPTION:
Study participants will receive either Henogen's adjuvanted hepatitis B vaccine or Aventis Pasteur's hepatitis B vaccine. The study involves a total of 4 visits and blood samples will taken at each of these visits.

ELIGIBILITY:
Inclusion criteria

* A male or female subject greater than or equal to 15 years of age at the time of study entry
* Written informed consent obtained from the subject/ from the parent or guardian of the subject.
* Seronegative for anti-HBc antibodies and for HBsAg at screening.
* Pre-dialysis patients, peritoneal dialysis patients or haemodialysis patients
* Documented evidence of previous hepatitis B vaccination with at least one full primary vaccination course of minimum four injections of licensed vaccine.
* The last dose should have been administered at least two months before the planned first dose of study vaccine in this study.
* Documented evidence of non-response to previous hepatitis B vaccination after at least one to maximum three months after the last vaccine dose.

Exclusion criteria

* Subject included on HN014/HBV-001 study. History of Hepatitis B infection Use of immunoglobulins within six months preceding the first study vaccination.
* Any confirmed or suspected human immunodeficiency virus (HIV) infection. Pregnant or lactating female

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 257 (Actual)
Dates: Start 2006-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Anti-HBs seroprotection rate | Month 2

SECONDARY OUTCOMES:
Anti-HBs Seroprotection rates for all subjects. | Months 0, 1 and 2
Anti-HBs Seropositivity rates for all subjects. | Months 0, 1 and 2
Percentage of subjects with anti-HBs antibody concentrations superior or equal to 100 mIU/ml for all subjects | Months 0, 1 and 2
Anti-HBs Geometric Mean Concentrations calculated for all subjects. | Months 0, 1 and 2
Occurrence and intensity of solicited local signs and symptoms, relationship to vaccination of solicited general signs and symptoms reported during the 4-day follow-up period after each vaccination and overall | Month 0, 1 and 2
Occurrence, intensity and relationship to vaccination of unsolicited signs and symptoms during the 31-day (Day 0 to Day 30) follow-up period after each vaccination and overall | Month 0, 1 and 2
Occurrence, intensity and relationship to vaccination of all serious adverse events (SAEs) up to Month 2 | Month 0 to 2

CONTACTS AND LOCATIONS:
Overall Officials: Christian Tielemans, MD, PhD, Principal Investigator — ULB Hôpital Erasme Département de Néphrologie
Locations (25):
- Belgium (13):
  - O.L.Vrouwziekenhuis Aalst, Aalst
  - RHMS La Madeleine ATH, Ath
  - RHMS Clinique Louis Caty Baudour, Baudour
  - Cliniques universitaires Saint Luc, Brussels
  - CHU Brugmann (site V Horta) Service de néphrologie, Brussels
  - ULB Hôpital Erasme Département de Néphrologie, Brussels
  - CHU Hôpital civil de, Charleroi
  - UZ AntwerpenDienst nefrologie, Edegem
  - UZ Gent, Ghent
  - CHU Tivoli, La Louvière
  - UZ Gasthuisberg Leuven Nierziekten, Leuven
  - CHU Andre VESALE, Montigny-le-Tilleul
  - RHMS TournayService de néphrologie, Tournai
- Czechia (6):
  - Clinic of Gerontology and MetabolismDepartment of NephrologyUniversity HospitalSokolska, Hradec Králové
  - Dept. of Heamodialysis Hospital JihlavaVrchlického, Jihlava
  - Dept. of NephrologyIII. Clinic of Internal DiseasesUniversity Hospital I.P.Pavlova, Olomouc
  - Infection Diseases and AIDS Treatment ClinicUniversity Hospital with Outpatient Clinic, Ostrava - Poruba
  - Fresenius Medical Care - DS, s.r.o.: PardubiceDialysis Unit Kyjevska, Pardubice
  - Fresenius Medical Care - DS, s.r.o.: SokolovDialysis Unit Slovenska, Sokolov
- Hungary (6):
  - University of Debrecen Medical and Science CenterI. Medical Clinic for Internal Diseases Nephrology Department, Debrecen
  - Markhot Ferenc County HospitalFresenius Dialysis Center Baktai, Eger
  - Vaszary Kolos HospitalFresenius Dialysis Center, Esztergom
  - Petz Aladár Teaching Hospital Vasvári, Győr
  - Hatvan Hospital Health Care ProviderFresenius Dialysis Center Hatvan ., Hatvan
  - Zala County HospitalII. Medical Department Nephrology Zrinyi, Zalaegerszeg